CLINICAL TRIAL: NCT03519204
Title: A Randomized, Multicenter, No-treatment Controlled Study of the Safety and Effectiveness of JUVÉDERM® VOLBELLA® With Lidocaine for Lip Enhancement in Chinese Adults
Brief Title: Safety and Effectiveness of JUVÉDERM® VOLBELLA® With Lidocaine for Lip Enhancement in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VOLBELLA-005
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2019-06-21 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Lip Enhancement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JUVÉDERM® VOLBELLA® XC with Lidocaine (Experimental): JUVÉDERM® VOLBELLA® XC with lidocaine injected into lips at Day 1. Participants were eligible to receive optional touch-up retreatment one month following initial treatment if applicable.
  Interventions: Device: JUVÉDERM® VOLBELLA® XC with Lidocaine
- No-treatment Control (Experimental): No-treatment was administered during control period. After 3 months, participants were eligible to receive treatment with JUVÉDERM® VOLBELLA® XC with lidocaine if applicable followed by an optional touch-up retreatment one month following initial treatment.
  Interventions: Device: JUVÉDERM® VOLBELLA® XC with Lidocaine; Other: No-treatment Control

INTERVENTIONS:
Device: JUVÉDERM® VOLBELLA® XC with Lidocaine — JUVÉDERM® VOLBELLA® XC with lidocaine injected into lips.
Other: No-treatment Control — No-treatment was administered.
  Arms: No-treatment Control

SUMMARY:
This study will evaluate the safety and effectiveness of VOLBELLA with Lidocaine injectable gel in Chinese adults seeking lip enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older with an overall baseline Lip Fullness Scale (LFS) score of minimal, mild or moderate on the 5-point LFS scale.
* Has the ability to follow study instructions and is likely to complete all required visits

Exclusion Criteria:

* Has had any facial procedures or trauma that may interfere with the study procedures and results
* Is on anti-coagulation therapy or other contraindicated treatments
* Has current cutaneous inflammatory or infectious processes or lesions in the mouth area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smita Chawla, Study Director — Allergan
Locations (5):
- China (5):
  - General Hospital of Southern Theatre Command, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - China-Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing

REFERENCES:
- [Derived] Li D, Gao Z, Sun J, Li Q, Jiang P, Zhang L, Chawla S. Safe and Effective Lip Enhancement with VYC-15L in Chinese Adults. Clin Cosmet Investig Dermatol. 2022 Nov 10;15:2427-2436. doi: 10.2147/CCID.S382194. eCollection 2022. PMID 36387967
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were randomized to the no-treatment control group but were treated in error on the day of randomization and were included in the treatment group for the Modified-intent-to-treat (mITT) population and the Safety population for analysis.
Period: Overall Study
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Started | 43 (3 control participants were treated in error; 29 participants received treatment after 3 months.) | 133
mITT Population | 33 | 130
Safety Population | 40 | 136
Completed | 30 | 118
Not Completed | 13 | 15
Not completed — Lost to Follow-up | 3 | 8
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Other Miscellaneous Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: mITT population included all participants who were randomized to study treatment (treatment group), received at least 1 study device treatment, and had baseline and at least 1 posttreatment assessment of primary variable, and who were randomized to no-treatment control group had baseline and at least 1 follow-up assessment of primary variable.
Groups:
- Total: Total of all reporting groups
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA® XC With Lidocaine | Total
Number analyzed (Participants) | 33 | 130 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (8.40) | 35.0 (9.83) | 35.0 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 127 | 158
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 33 | 130 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 33 | 130 | 163
Lip Fullness Scale (LFS) Score as Assessed by Evaluating Investigator (EI) [Count of Participants; unit: Participants] — The investigator assessed the participant's lip fullness using a 5-point scale where: 0=Minimal (Flat or nearly flat contour, minimal red lip show), 1=Mild (Some red lip show; no lower lip pout), 2=Moderate (Moderate red lip show with slight lower lip pout), 3=Marked (Significant red lip show and lower lip pout), and 4=Very Marked (Very significant red lip show, lower lip pout, and upper lip pout). Population: mITT population included all participants who were randomized to study treatment (treatment group), received at least 1 study device treatment, and had baseline and at least 1 posttreatment assessment of primary variable, and who were randomized to no-treatment control group had baseline and at least 1 follow-up assessment of primary variable.
  Participants
    Minimal | 1 | 7 | 8
    Mild | 16 | 59 | 75
    Moderate | 16 | 63 | 79
    Marked | 0 | 1 | 1
    Very Marked | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥1-point Increase (Improvement) on the Evaluating Investigator's (EI's) Assessed 5-point Lip Fullness Scale (LFS)
Description: The investigator assessed the participant's lip fullness using the 5-point LFS where: 0=Minimal (Flat or nearly flat contour, minimal red lip show), 1=Mild (Some red lip show; no lower lip pout), 2=Moderate (Moderate red lip show with slight lower lip pout), 3=Marked (Significant red lip show and lower lip pout), and 4=Very Marked (Very significant red lip show, lower lip pout, and upper lip pout). Improvement was defined as a ≥1-point increase in fullness from Baseline. Number analyzed is the number of participants with data available for analysis at Baseline and Month 3.
Time Frame: Baseline to Month 3 Post Last Treatment (JUVÉDERM® VOLBELLA® XC with Lidocaine arm) or Month 3 Post Randomization (No-treatment Control arm)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- No-treatment Control: No-treatment was administered during control period.
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 29 | 118
percentage of participants | 0 [0.0 to 11.9] | 84.7 [77.0 to 90.7]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLBELLA® XC With Lidocaine; Test type: Superiority; p < 0.0001, Fisher Exact — P-value was based on 2-sided Fisher's exact test comparing responder rate between treatment group and no-treated control group; Responder Rate Difference = 84.7, 95% CI 2-sided [68.2 to 94.2]

2. Secondary Outcome: Percentage of Participants With a ≥1-point Increase (Improvement) Based on the Participant's Assessed 5-point LFS
Description: Lip fullness was assessed by the participant using the 5-point LFS where: 0=Minimal (Flat or nearly flat contour, minimal red lip show), 1=Mild (Some red lip show; no lower lip pout), 2=Moderate (Moderate red lip show with slight lower lip pout), 3=Marked (Significant red lip show and lower lip pout), and 4=Very Marked (Very significant red lip show, lower lip pout, and upper lip pout). Improvement was defined as a ≥1-point increase in fullness from Baseline. Number analyzed is the number of participants with data available for analysis at Baseline and Month 3.
Time Frame: Baseline to Month 3 Post Treatment
Population: mITT population included all participants who were randomized to study treatment (treatment group), received at least 1 study device treatment, and had baseline and at least 1 posttreatment assessment of the primary variable. As per protocol, analysis for this Outcome Measure was for the Treatment arm only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 117
percentage of participants | 65.0 [55.6 to 73.5]

3. Secondary Outcome: Change From Baseline in Overall Lip Volume
Description: Overall lip volume was measured by 3-dimensional (3D) photography images. A positive change from Baseline indicates improvement. Number analyzed is the number of participants with data available for analysis at Baseline and Month 3.
Time Frame: Baseline to Month 3 Post Treatment ( JUVÉDERM® VOLBELLA® XC with Lidocaine arm) or Month 3 Post Randomization (No-treatment Control arm)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: cubic centimeters (cc)
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 27 | 108
cubic centimeters (cc) | 0.03990 [-2.2055 to 0.5676] | 0.45150 [-0.8456 to 1.9478]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLBELLA® XC With Lidocaine; Test type: Superiority; p < 0.0001, Wilcoxon Rank-sum Test — P-value was computed using Wilcoxon test with normal approximation; Median Difference = 0.55800, 95% CI 2-sided [0.34470 to 0.77390], Standard Error of Mean 0.109492 — The median difference (the location shift) and its 95% CI were computed using Hodges-Lehmann estimation associated with Wilcoxon statistics

4. Secondary Outcome: Percentage Change From Baseline in Lip Surface Area
Description: Lips surface area was measured by 3D photography images. A positive percentage change from Baseline indicates improvement. Number analyzed is the number of participants with data available for analysis at Baseline and Month 3.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percentage change in lip surface area
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 29 | 113
percentage change in lip surface area | -0.11 [-21.5 to 20.1] | 12.16 [-9.5 to 76.9]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLBELLA® XC With Lidocaine; Test type: Superiority; p < 0.0001, Wilcoxon Rank-sum Test — P-value was computed using Wilcoxon test with normal approximation; Median Difference = 13.04, 95% CI 2-sided [8.861 to 17.180], Standard Error of Mean 2.122 — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Procedural Pain Score
Description: Procedural pain (pain during injection) was evaluated by the participant using an 11-point scale, where: 0=No pain to 10=Worst pain imaginable. Participants recorded procedural pain in safety diary for 30 days after initial treatment. Number analyzed is the number of participants with safety diary data available for analysis.
Time Frame: Up to 30 days after initial treatment with JUVÉDERM® VOLBELLA® XC with Lidocaine
Population: Safety population included all participants randomized to the treatment group who received at least 1 study treatment and all participants randomized to the control group, as treated. Analysis excludes 11 participants in the No-treatment Control group who did not receive JUVÉDERM® VOLBELLA®.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treated Control: No-treatment was administered during control period. After 3 months, participants received treatment with JUVÉDERM® VOLBELLA® XC with lidocaine if applicable followed by an optional touch-up retreatment one month following initial treatment.
Arm/Group | Treated Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 29 | 136
score on a scale | 2.6 (1.86) | 2.6 (1.69)

6. Secondary Outcome: Number of Participants With Injection Site Responses (ISRs)
Description: ISRs were recorded by the participant in a safety diary for 30 days after each treatment and were summarized by treatment (initial and touch-up). ISRs were defined as redness, pain after injection, tenderness to touch, firmness, swelling, lumps/bumps, bruising, itching and discoloration. Number analyzed is the number of participants with safety diary data available for analysis.
Time Frame: Up to 30 days after each treatment with JUVÉDERM® VOLBELLA® XC with Lidocaine
Population: Safety population included all participants randomized to the treatment group who received at least 1 study treatment and all participants randomized to the control group, as treated. Analysis excludes 11 participants in the No-treatment Control group who did not receive JUVÉDERM® VOLBELLA® XC with Lidocaine.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Control | JUVÉDERM® VOLBELLA® XC With Lidocaine
Number analyzed (Participants) | 29 | 136
Participants
  Initial Treatment: number analyzed (Participants) | 28 | 130
  Initial Treatment | 26 | 123
  Touch-up Treatment: number analyzed (Participants) | 6 | 32
  Touch-up Treatment | 6 | 26

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) is any untoward medical occurrence in a patient or a participant using an investigational drug, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A TEAE is an AE that occurred after receiving the first dose of study device or study injection or an AE present prior to first dose but increased in severity during the Treatment Period.
Time Frame: Baseline to Month 12 Post Treatment
Population: Safety population included all participants randomized to the treatment group who received at least 1 study treatment and all participants randomized to the control group, as treated.
Measure: Count of Participants; unit: Participants
Groups:
- No-treatment Control (Control Period): No-treatment was administered during control period.
- JUVÉDERM® VOLBELLA® XC With Lidocaine (All Treated): JUVÉDERM® VOLBELLA® XC with lidocaine injected into lips at Day 1. Participants were eligible to receive optional touch-up retreatment one month following initial treatment if applicable.
  Includes 29 participants in the No-treatment Control arm who received treatment with JUVÉDERM® VOLBELLA® XC with Lidocaine injected into lips after 3 months.
Arm/Group | No-treatment Control (Control Period) | JUVÉDERM® VOLBELLA® XC With Lidocaine (All Treated)
Number analyzed (Participants) | 40 | 165
Participants | 3 | 74

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12 Post Treatment
Description: Safety population included all participants randomized to the treatment group who received at least 1 study treatment and all participants randomized to the control group, as treated. 29 participants in the No-treatment Control arm received JUVÉDERM® VOLBELLA® XC with Lidocaine after 3 months and are included in the JUVÉDERM® VOLBELLA® XC with Lidocaine arm.
Arm/Group | No-treatment Control (Control Period) | JUVÉDERM® VOLBELLA® XC With Lidocaine (All Treated)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/40 | 5/165
Other Adverse Events (participants affected / at risk) | 1/40 | 40/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (Control Period) (N=40) | JUVÉDERM® VOLBELLA® XC With Lidocaine (All Treated) (N=165)
Injection site ischaemia (General disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (Control Period) (N=40) | JUVÉDERM® VOLBELLA® XC With Lidocaine (All Treated) (N=165)
Injection site induration (General disorders) | 0 | 24
Injection site mass (General disorders) | 0 | 10
Upper respiratory tract infection (Infections and infestations) | 1 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03519204/SAP_000.pdf
  • Study Protocol (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03519204/Prot_001.pdf